CLINICAL TRIAL: NCT03743220
Title: Construction and Validation of a Simplified Provocation Tests for the Diagnosis of Non Steroidal Anti-inflammatory Drugs (NSAID) Hypersensitivity
Brief Title: Drug Provocation Test (DPT) to Non Steroidal Anti-inflammatory Drugs (NSAID)
Acronym: NSAID
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0433
Record Dates: First submitted 2018-11-13; First posted 2018-11-16 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Drug Hypersensitivity
Keywords: Drug Hypersensitivity Reaction; Drug Provocation Test; Non steroidal Anti Inflammatory drugs; Reactive Doses; Reactive Times
MeSH Terms: conditions — Drug Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background : Non steroidal anti-inflammatory drugs are responsible for 25% of reported adverse drug events which include immunological and non-immunological hypersensitivity reactions. NSAIDs have been reported to be the second most common cause of drug-induced hypersensitivity reaction (DHR). They are almost mandatory in a human life and therefore, the drug allergy work-up goes up until a DPT in order to confirm or rule out the diagnosis.

Objective: Detect eliciting dose thresholds during NSAIDs DPT in order to suggest optimal step doses and to describe subgroups at higher risk during the DPT

Methods:This retrospective study, using the survival analysis, comprised all patients who attended the allergy service of the UH of Montpellier from 1997 till 2017 with a clinical history related to NSAIDs DHR, who underwent NDAIDs DPT that turned positive and who gave their consent to be included in the study . The Patients are selected from the Drug Allergy & Hypersensitivity Database (DAHD).

DETAILED DESCRIPTION:
DHRs to NSAIDs may be induced by both specific immunological mechanisms and mechanisms not based on immunological recognition (cross-hypersensitivity reactions [CRs]) .They are almost mandatory in a human life and therefore, the drug allergy work-up goes up until a DPT in order to confirm or rule out the diagnosis. Although the overall prevalence of NSAID hypersensitivity has been reported between 0.6 and 7% of the general population .

The NSAIDs-induced hypersensitivity reactions involve different mechanisms and present a wide range of clinical manifestations from anaphylaxis or severe bronchospasm developing within minutes after drug ingestion to non-immediate responses appearing after days and weeks This data-driven approach in designing the DPT protocol is the second step in improving DPT standardization, after BL antibiotics.

ELIGIBILITY:
Inclusion criteria:

- Patients with one or more positives DPT to NSAIDs

Exclusion criteria:

- Patients refusing to take part in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient consulting in our allergy unit for a suspicion of drug hypersensitivity to non steroidal anti inflammatory drug (s) and who underwent DPT.
Sampling Method: Non-Probability Sample
Enrollment: 311 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Detect eliciting dose thresholds during NSAIDs DPT optimal step doses | 1 day
  The DPT was considered positive if objective signs occurred during NSAIDs administration. The reactive dose (RD) was calculated from the total cumulative dose (mg) reached when the DPT was considered positive

SECONDARY OUTCOMES:
Describe subgroups at higher risk during the DPT | 1 day
  Identifying the independent variables (predictive factors), using the multivariate linear regression method, that remains significantly associated with a positive NSAIDs DPT

CONTACTS AND LOCATIONS:
Overall Officials: Pascal DEMOLY, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No